CLINICAL TRIAL: NCT04030026
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled, Two-Treatment, Two-Period Crossover Efficacy and Safety Study in Idiopathic Pulmonary Fibrosis (IPF) With Nalbuphine ER Tablets for the Treatment of Cough
Brief Title: A Study of Nalbuphine (Extended Release) ER in Idiopathic Pulmonary Fibrosis (IPF) for Treatment of Cough
Acronym: CANAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR12; 2018-004744-31 (EudraCT Number)
Record Dates: First submitted 2019-07-11; First posted 2019-07-23 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Nalbuphine; Cough; Idiopathic Pulmonary Fibrosis; Pharmacokinetics
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough | interventions — Nalbuphine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, 2-Treatment, 2-Period Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NAL ER then placebo (Experimental): Participants received NAL ER in treatment period 1 at dose 27 mg once daily (QD) to 54 mg twice daily (BID) over a 5-day period and then maintained at 54 mg BID for 4 days. Dose was increased to 108 mg BID for 1 week then to 162 mg BID for 6 days, followed by placebo matching NAL ER for 3 weeks in treatment period 2. Both the treatment periods were separated by 2 weeks of washout period.
  Interventions: Drug: NAL ER; Drug: Placebo
- Placebo then NAL ER (Experimental): Participants received placebo matching NAL ER for 3 weeks in treatment period 1 followed by NAL ER in treatment period 2 at dose 27 mg QD to 54 mg BID over a 5-day period and then maintained at 54 mg BID for 4 days. Dose was increased to 108 mg BID for 1 week then to 162 mg BID for 6 days. Both the treatment periods were separated by 2 weeks of washout period.
  Interventions: Drug: NAL ER; Drug: Placebo

INTERVENTIONS:
Drug: NAL ER — Participants received NAL ER 27 mg QD, 27 mg BID, 54 mg BID, 108 mg BID, 162 mg BID.
  Other Names: Nalbuphine
Drug: Placebo — Participants received Placebo tablet (matching NAL ER ).
  Other Names: Placebo matched to NAL ER

SUMMARY:
To evaluate the safety and tolerability of nalbuphine ER tablets in the study population and to evaluate the effect of NAL ER tablets on the mean daytime cough frequency (coughs per hour) at Day 22 (dose 162 mg BID) as compared to placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals diagnosed with Idiopathic Pulmonary Fibrosis
2. Chronic cough > 8 weeks.
3. Daytime cough severity score ≥ 4 on Cough Severity Numerical Rating Scale at screening.

Exclusion Criteria:

1. The following conditions are excluded:

   1. Interstitial lung disease (ILD) known to be caused by domestic and occupational environmental exposures.
   2. Interstitial lung disease (ILD) known to be caused by connective tissue disease.
   3. Interstitial lung disease (ILD) known to be caused by drug related toxicity.

      2. Currently on continuous oxygen therapy.

      3. History of substance abuse that, as determined by the Investigator, may interfere with the conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sciascia, Study Director — Trevi Therapeutics, Inc
Locations (11):
- United Kingdom (11):
  - 09, Cambridge
  - 08, Cottingham
  - 17, Dundee
  - 13, Edinburgh
  - 04, London
  - 01, London
  - 02, Manchester
  - 10, Newcastle upon Tyne
  - 06, Nottingham
  - 14, Oxford
  - 03, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maher TM, Avram C, Bortey E, Hart SP, Hirani N, Molyneux PL, Porter JC, Smith JA, Sciascia T. Nalbuphine Tablets for Cough in Patients with Idiopathic Pulmonary Fibrosis. NEJM Evid. 2023 Aug;2(8):EVIDoa2300083. doi: 10.1056/EVIDoa2300083. Epub 2023 May 22. PMID 38320144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 11 sites in the United Kingdom from 29 October 2019 to 27 May 2022.
Pre-assignment Details: A total of 56 participants were screened from whom 42 participants were enrolled and randomized to receive treatment in this study.
Groups:
- First NAL ER Then Placebo: Participants received NAL ER in treatment period 1 at dose 27 mg once daily (QD) to 54 mg twice daily (BID) over a 5-day period and then maintained at 54 mg BID for 4 days. Dose was increased to 108 mg BID for 1 week then to 162 mg BID for 6 days, followed by placebo for 3 weeks in treatment period 2. Both the treatment periods were separated by 2 weeks of washout period.
- First Placebo Then NAL ER: Participants received placebo for 3 weeks in treatment period 1 followed by NAL ER in treatment period 2 at dose 27 mg QD to 54 mg BID over a 5-day period and then maintained at 54 mg BID for 4 days. Dose was increased to 108 mg BID for 1 week then to 162 mg BID for 6 days. Both the treatment periods were separated by 2 weeks of washout period.
Period: Treatment Period 1 (22 Days)
Arm/Group | First NAL ER Then Placebo | First Placebo Then NAL ER
Started | 21 | 21
Safety Analysis Set (Safety Analysis Set (SAS) included all randomized participants who had received at least 1 dose of the investigational product (IP).) | 20 | 21
Completed | 19 | 19
Not Completed | 2 | 2
Not completed — COVID-19 pandemic restrictions | 0 | 1
Not completed — Withdrawal by Participant | 1 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Physician Decision | 1 | 0
Period: Treatment Period 2 (22 Days)
Arm/Group | First NAL ER Then Placebo | First Placebo Then NAL ER
Started | 19 | 19
Completed | 18 | 10
Not Completed | 1 | 9
Not completed — Adverse Event | 0 | 6
Not completed — COVID-19 pandemic restrictions | 1 | 1
Not completed — Withdrawal by Participant | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized analysis set included all participants who were randomized.
Groups:
- First NAL ER Then Placebo: Participants received NAL ER in treatment period 1 at dose 27 mg QD to 54 mg BID over a 5-day period and then maintained at 54 mg BID for 4 days. Dose was increased to 108 mg BID for 1 week then to 162 mg BID for 6 days, followed by placebo for 3 weeks in treatment period 2. Both the treatment periods were separated by 2 weeks of washout period.
- Total: Total of all reporting groups
Arm/Group | First NAL ER Then Placebo | First Placebo Then NAL ER | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Customized [Number; unit: years]
  18-64 years | 3 | 1 | 4
  65-85 years | 18 | 19 | 37
  85 years and above | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 19 | 17 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 4
  White | 20 | 18 | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 20 | 20 | 40
  Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A TEAE was defined as any AE that occurs after the first dose of study drug. TEAEs included both serious and non-serious TEAEs.
Time Frame: Up to Day 72
Population: SAS included all randomized participants who had received at least 1 dose of the IP. 3 participants did not receive at least one dose of NAL ER but received placebo and 1 participant did not receive at least one dose of placebo but received NAL ER treatment. Data was summarized under actual treatment received (NAL ER or placebo) independently whether this was received in Treatment Period 1 or 2 (participants who received both treatments are counted in both NAL ER and placebo columns).
Measure: Count of Participants; unit: Participants
Groups:
- NAL ER: Participants received NAL ER 27 mg QD to 54 mg BID over a 5-day period, and then maintained at 54 mg BID for 4 days. Dose was increased to 108 mg BID for 1 week followed by 162 mg, BID for 6 days in treatment period 1 or 2 of the study.
- Placebo: Participants received placebo for 3 weeks through treatment period 1 or 2 of the study.
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 40
Participants | 35 | 26

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: The clinical laboratory parameters included the urinalysis, hematology, serum chemistry, coagulation and liver function parameters. Clinical significance was determined by the investigator.
Time Frame: Up to Day 72
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 40
Participants
  Urinalysis | 0 | 0
  Hematology | 1 | 0
  Serum Chemistry | 1 | 1
  Coagulation | 0 | 1
  Liver Function Parameters | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Sign Parameters
Description: Vital signs measurements included blood pressure, heart rate, and respiration rate, body temperature, pulse oximetry, and weight. Clinical significance was determined by the investigator.
Time Frame: Up to Day 72
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 40
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination Parameters
Description: Physical examination included examination of the following body systems: general appearance, eyes, ears, nose, throat, head and neck, chest and lungs, cardiovascular, abdomen, musculoskeletal, lymphatic, dermatological, neurological, and extremities. Clinical significance was determined by the investigator.
Time Frame: Up to Day 72
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 40
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECG)
Description: Changes in ECG data such as heart rate, rhythm, and other clinically significant abnormalities (left ventricular hypertrophy, pathological Q-waves) were measured. Clinical significance was determined by the investigator.
Time Frame: Up to Day 72
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 40
Participants | 1 | 1

6. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Day 21
Description: Spirometry was used to assess FVC. It was used to assess pulmonary breathing mechanics.
Time Frame: Baseline, Day 21
Population: Participants in SAS were analyzed.3 participants did not receive at least 1 dose of NAL ER but received placebo and 1 participant did not receive at least 1 dose of placebo but received NAL ER treatment. Data was summarized under actual treatment received (NAL ER or placebo) independently whether in Treatment Period 1 or 2 (participants who received both treatments are counted in both NAL ER and placebo columns).Overall number of participants analyzed'=participants who were evaluable for the OM.
Measure: Mean (Standard Deviation); unit: litre(s)
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 28 | 35
litre(s) | -2.3 (5.58) | -1.0 (5.56)

7. Primary Outcome: Subjective Opiate Withdrawal (SOWS) Total Raw Score
Description: The SOWS is a self-administered scale for grading opioid withdrawal symptoms and was collected via the study issued e-diary. It consisted of 16 symptoms related to how the participant felt. Each symptom was scored between 0 to 4. The total score ranges between 0 to 64, higher score indicates more severe symptoms.
Time Frame: Up to Day 72
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 36 | 38
score on a scale | 4.7055 (5.0019) | 2.4082 (3.5561)

8. Primary Outcome: Daytime Cough Frequency at Baseline
Description: Daytime cough was defined as cough that occurs between the time that the participant is a wake in the 24 hours after the digital cough monitor was applied for use. Assessment was done using objective digital cough monitoring. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: At Baseline
Population: Full Analysis Set (FAS) included all randomized participants who had received at least single dose of the study medication and provided study baseline and at least one post -baseline primary efficacy variable assessment during the treatment Period.
Measure: Mean (Standard Deviation); unit: coughs per hour
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 38
coughs per hour | 27.99 (23.704) | 27.99 (23.704)

9. Primary Outcome: Percent Change From Baseline in Daytime Cough Frequency at Day 22
Description: Daytime cough was defined as cough that occurs between the time that the participant is a wake in the 24 hours after the digital cough monitor was applied for use. Assessment was done using objective digital cough monitoring. Percent change in daytime cough frequency (coughs per hour) from baseline was assessed. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Day 22
Population: FAS included all randomized participants who had received at least single dose of the study medication and provided study baseline and at least one post -baseline primary efficacy variable assessment during the treatment Period. 'Overall number of participants analyzed' included those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 29 | 37
percent change | -75.11 [-82.655 to -67.567] | -22.62 [-42.531 to 2.715]
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects model — Mixed-effects model: unstructured, heterogeneous toeplitz and autoregressive covariance matrices. Dependent variable: change from baseline in log-transformed scale of Daytime Cough Frequency. Fixed effects: sequence (arm), period and treatment; Geometric Mean Ratio = 0.32, 95% CI 2-sided [0.208 to 0.431]

10. Secondary Outcome: Change From Baseline in Daytime Cough Frequency at Day 22
Description: Daytime cough was defined as cough that occurs between the time that the participant wakes up and the time that the participant goes to bed. Assessment was done using objective digital cough monitoring. The change in daytime cough frequency (coughs per hour) from baseline was assessed. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Day 22
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: coughs per hour
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 29 | 37
coughs per hour | -19.386 (19.5688) | -6.264 (12.4006)

11. Secondary Outcome: Percent Change From Baseline in 24-Hour Cough Frequency at Day 22
Description: Percent change in 24-hour (combined daytime and nighttime) cough frequency (coughs per hour) from baseline was assessed. Assessment was done using objective digital cough monitoring. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Day 22
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 29 | 37
percent change | -76.10 [-83.133 to -69.075] | -25.29 [-43.894 to -6.690]
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects model — [p-value comment as in outcome 9, analysis 1]; Geometric Mean Ratio = 0.32, 95% CI 2-sided [0.208 to 0.431]

12. Secondary Outcome: Percent Change From Baseline in Nighttime Cough Frequency at Day 22
Description: Nighttime cough frequency was intended as the average coughs per hour while the participant was flagged as being asleep. Assessment was done using objective digital cough monitoring. Percent change in cough frequency (coughs per hour) from baseline was assessed. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Day 22
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 29 | 37
percent change | -62.27 [-79.588 to -44.957] | -20.30 [-51.391 to 10.783]
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p = 0.0087, Mixed-effects model — [p-value comment as in outcome 9, analysis 1]; Geometric Mean Ratio = 0.47, 95% CI 2-sided [0.230 to 0.717]

13. Secondary Outcome: Mean Change From Baseline in the Evaluating Respiratory Symptoms (E-RS) Diary Cough Subscale at Days 9, 16, and 22
Description: E-RS daily diary instrument has four separate respiratory symptom domain scales which is a valid, reliable and sensitive measure of four distinct respiratory symptoms. The four domain scales that included cough [E-RS item 2- How often did you cough today?;score range 0 (not at all)-4 (almost constantly)], and other items such as breathlessness [score 0(not at all)-23(severe symptoms)], sputum [0(not at all)-8(severe symptoms)], and chest symptoms [0(not at all)-12(severe symptoms)]. The raw totals for the E-RS score and for each of the subscales were converted to a scale range of 0 to 100 (least symptomatic to most symptomatic). A higher score on the scale indicates a more severe grade to the symptom. Negative score indicates improvement in the symptom. The mean change from baseline in the E-RS diary cough scores was assessed. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Days 9, 16, and 22
Population: FAS included all randomized participants who had received at least single dose of the study medication and provided study baseline and at least one post -baseline primary efficacy variable assessment during the treatment Period. 'Number analyzed' indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 38
score on a scale
  Change at Day 9: number analyzed (Participants) | 32 | 38
  Change at Day 9 | -0.7 (0.77) | -0.1 (0.70)
  Change at Day 16: number analyzed (Participants) | 30 | 38
  Change at Day 16 | -0.9 (0.82) | -0.2 (0.59)
  Change at Day 22: number analyzed (Participants) | 27 | 32
  Change at Day 22 | -1.0 (0.94) | -0.2 (0.85)
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Change from baseline at Day 9; Test type: Superiority; p = 0.0014, Student's T-test — Student's T-test was used to evaluate if the difference in mean change from baseline is different between planned treatments (NAL ER vs placebo)
Statistical Analysis 2: Comparison: NAL ER vs Placebo; Change from baseline at Day 16; Test type: Superiority; p = 0.0001, Student's T-test — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: NAL ER vs Placebo; Change from baseline at Day 22; Test type: Superiority; p = 0.001, Student's T-test — [p-value comment as in outcome 13, analysis 1]

14. Secondary Outcome: Mean Change From Baseline in E-RS Breathlessness Score at Days 9, 16, and 22
Description: E-RS daily diary instrument has four separate respiratory symptom domain scales which is a valid, reliable and sensitive measure of four distinct respiratory symptoms. The four domain scales included breathlessness [E-RS items 7 (were you breathless today), 8 (how breathless were you today), 9 (breathlessness doing personal care activities),10 (breathlessness doing indoor activities) & 11 (breathlessness doing outdoor activities); score =0: not at all) - 23: almost constantly]. Other items were cough (0: not at all-4: severe), sputum (0: not at all-8: severe), and chest symptoms (0: not at all)-12: severe symptoms). The raw totals for the E-RS score and for subscales were converted to a scale of 0 to 100 (least to most symptoms). Higher score=more severe grade to the symptom. Negative score=improvement in symptom. The mean change from baseline was assessed. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Days 9, 16, and 22
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 38
score on a scale
  Change at Day 9: number analyzed (Participants) | 32 | 38
  Change at Day 9 | -0.5 (2.68) | 1.1 (2.74)
  Change at Day 16: number analyzed (Participants) | 30 | 38
  Change at Day 16 | 0.0 (2.30) | 1.2 (2.26)
  Change at Day 22: number analyzed (Participants) | 27 | 32
  Change at Day 22 | 0.1 (2.45) | 0.8 (2.43)
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Change from baseline at Day 9; Test type: Superiority; p = 0.0198, Student's T-test — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: NAL ER vs Placebo; Change from baseline at Day 16; Test type: Superiority; p = 0.0374, Student's T-test — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: NAL ER vs Placebo; Change from baseline at Day 22; Test type: Superiority; p = 0.2982, Student's T-test — [p-value comment as in outcome 13, analysis 1]

15. Secondary Outcome: Mean Change From Baseline in the Cough Severity Numerical Rating Scale (NRS) at Days 8, 15, and 21
Description: The Cough Severity NRS instrument is a single-dimension 11-point Likert scale ranging from 0 (no cough) to 10 (worst possible cough). Negative score indicates improvement in the symptoms. Participants completed the cough numerical severity rating via the study specific e-diary. The mean change from baseline in the Cough Severity Numerical Rating Scale was assessed. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Days 8, 15, and 21
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 38
score on a scale
  Change at Day 8: number analyzed (Participants) | 27 | 38
  Change at Day 8 | -1.7 (1.98) | -0.4 (1.54)
  Change at Day 15: number analyzed (Participants) | 29 | 37
  Change at Day 15 | -2.7 (1.75) | -0.6 (1.74)
  Change at Day 21: number analyzed (Participants) | 27 | 33
  Change at Day 21 | -2.5 (2.19) | -0.3 (1.85)
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Change from baseline at Day 8; Test type: Superiority; p = 0.0054, Student's T-test — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: NAL ER vs Placebo; Change from baseline at Day 15; Test type: Superiority; p < 0.0001, Student's T-test — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: NAL ER vs Placebo; Change from baseline at Day 21; Test type: Superiority; p = 0.0001, Student's T-test — [p-value comment as in outcome 13, analysis 1]

16. Secondary Outcome: Mean Change From Baseline in the 14-item EXAcerbation of Chronic Pulmonary Disease Tool (EXACT) v1.1 e-Diary Tool Total Score at Days 9, 16, and 22
Description: The EXACT tool is a 14-item Daily Diary Tool Patient-reported outcome (PRO) instrument that was developed to quantify and measure exacerbations of chronic obstructive pulmonary disease (COPD). It provides a total score and subscale scores for breathlessness, cough and sputum, and chest symptoms. The 14 items have interval-level scale ranging between 0 to 100. The total score of each domain of breathlessness, cough and sputum, and chest symptoms ranges from 0 to 100. A higher score indicates a more severe condition. Negative score indicated improvement in the symptoms. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Days 9, 16, and 22
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 38 | 38
score on a scale
  Change at Day 9: number analyzed (Participants) | 32 | 38
  Change at Day 9 | -2.0 (5.63) | 1.6 (5.55)
  Change at Day 16: number analyzed (Participants) | 30 | 38
  Change at Day 16 | -1.8 (4.89) | 1.9 (5.46)
  Change at Day 22: number analyzed (Participants) | 27 | 32
  Change at Day 22 | -1.6 (5.92) | 0.6 (5.76)
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Change from baseline at Day 9; Test type: Superiority; p = 0.0107, Student's T-test — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: NAL ER vs Placebo; Change for baseline at Day 16; Test type: Superiority; p = 0.0051, Student's T-test — [p-value comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: NAL ER vs Placebo; Change from baseline at Day 22; Test type: Superiority; p = 0.1513, Student's T-test — [p-value comment as in outcome 13, analysis 1]

17. Secondary Outcome: Mean Change From Baseline in the Patient Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 Fatigue Short Form 7a Scale Total Score at Day 21
Description: The PROMIS Fatigue Short Form 7a is a self-administered Likert-type rating 5-point scale of 7 questions that assess tiredness, exhaustion, energy, fatigue limit, tiredness to think, tiredness impact on hygiene and impact on ability to exercise strenuously over the past 7 days. It consisted of 7 items with each item was scored between 1 to 5. The total score could range between 1 to 35, higher score indicates more severe symptoms. Baseline was defined as the last available assessment prior to the first Treatment Period 1 IP intake.
Time Frame: Baseline, Day 21
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 24 | 30
score on a scale | 0.9 (3.98) | 0.0 (2.98)
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p = 0.3601, Student's T-test — [p-value comment as in outcome 13, analysis 1]

18. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Over Time Measured at Day 21
Description: The CGI-C is a one-item measure evaluating change from the initiation of treatment on a 7-point scale. It provides an overall clinician-determined summary measure that takes into account all available information, including knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. The total score ranges between 0 (very much improved) to 7 (very much worse). The lower scores indicate an improvement in respiratory symptoms.
Time Frame: At Day 21
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 29 | 36
score on a scale | 3.0 (1.50) | 3.9 (0.91)

ADVERSE EVENTS:
Time Frame: Up to Day 72
Description: All-cause mortality:All randomized participants.Adverse events:SAS=all randomized participants who received at least 1 dose of IP.3 participants did not receive at least 1 dose of NAL ER but received placebo,1 participant did not receive at least 1 dose of placebo but received NAL ER treatment.Data was summarized under actual treatment received independently whether this was received in Treatment Period 1/2(participants who received both treatments are counted in both NAL ER,placebo columns).
Arm/Group | NAL ER | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/38 | 1/40
Other Adverse Events (participants affected / at risk) | 35/38 | 26/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NAL ER (N=38) | Placebo (N=40)
Urosepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NAL ER (N=38) | Placebo (N=40)
Dizziness (Nervous system disorders) | 10 | 0
Somnolence (Nervous system disorders) | 9 | 1
Headache (Nervous system disorders) | 5 | 5
Lethargy (Nervous system disorders) | 3 | 2
Fatigue (General disorders) | 12 | 3
Nausea (Gastrointestinal disorders) | 16 | 0
Constipation (Gastrointestinal disorders) | 11 | 2
Vomiting (Gastrointestinal disorders) | 7 | 5
Dry Mouth (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Anxiety (Psychiatric disorders) | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT04030026/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT04030026/SAP_001.pdf